CLINICAL TRIAL: NCT00665041
Title: A Randomised, Double-blind, Parallel Groups, Placebo-controlled, Single-centre Pilot Study Assessing the Tolerability of Quinagolide in a Dose-titration Regimen in Oocyte Donors at Risk of Developing Ovarian Hyperstimulation Syndrome
Brief Title: Tolerability of Quinagolide in a Dose-titration Regimen in Oocyte Donors at Risk of Developing Ovarian Hyperstimulation Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr Antonio Pellicer, Instituto Valenciano de Infertilidad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VLC-CB-090108-001; NCT00742651 (obsolete NCT alias)
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — quinagolide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PR1 (Experimental)
  Interventions: Drug: Quinagolide
- PL1 (Placebo Comparator)
  Interventions: Drug: Quinagolide

INTERVENTIONS:
Drug: Quinagolide — • Quinagolide 200 μg/day (dose titration from 50 μg/day to 100 μg/day to 200 μg/day), oral. Quinagolida tablets, 50 mcg.
  placebo, oral.

SUMMARY:
Assess the tolerability of quinagolide 200 μg/day in a dose-titration regimen in oocyte donors undergoing controlled ovarian hyperstimulation and at risk of developing OHSS Secondary Objectives

Estimate the effects of a quinagolide dose-titration regimen compared to placebo in peritoneal fluid accumulation, incidence of ascites, OHSS symptoms and clinical laboratory parameters of haemoconcentration

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form, prior to screening evaluations
2. In good physical and mental health
3. Pre-menopausal females between the ages of 21-34 years (both inclusive) at the time of randomisation
4. Body mass index (BMI) between 18 and 29 kg/m2 (both inclusive)
5. Oocyte donor currently undergoing a controlled ovarian hyperstimulation cycle for assisted reproductive technologies (ART)
6. Antral follicle count ≥ 20

Exclusion Criteria:

1. Any exclusion criteria for oocyte donation
2. Known clinically significant systemic disease (e.g., insulin dependent diabetes)
3. Known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) which can compromise participation in the study
4. Undiagnosed vaginal bleeding
5. Known tumours of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus
6. Malformations of the sexual organs incompatible with pregnancy
7. Positive pregnancy test prior to start of stimulation
8. Treatment with other dopamine agonists (ATC code N04BC) or dopamine antagonists (ATC code N05A) within 2 months prior to randomisation
9. Treatment with any hormonal therapy (except for thyroid medication and oral contraceptives and except that routinely used as part of the controlled ovarian hyperstimulation cycle), anti-psychotics (ATC code N05A), anti-depressants (ATC code N06), anxiolytics (ATC code N05B), hypnotics and sedatives (ATC code N05C) or continuous use of prostaglandin inhibitors (non-steroid anti-inflammatory drugs (NSAIDs), including aspirin) within 2 weeks prior to randomisation
10. Known hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
11. Known history of psychotic disorders
12. Hypotension, orthostatic hypotension or recurrent syncope within 6 months prior to randomisation
13. Ongoing treatment of hypertension
14. Known previous poor tolerability to dopamine agonists
15. Known impaired hepatic or renal function
16. Current or past (12 months prior to randomisation) abuse of alcohol or drugs, and/or current (last month prior to randomisation) use of alcohol (more than 14 units per week)
17. Current or past (3 months prior to randomisation) smoking habit of more than 20 cigarettes per day
18. History of chemotherapy (except for gestational conditions) or radiotherapy
19. Use of any investigational drug during 3 months prior to randomisation
20. Previous participation in the study
21. Hypersensitivity to the active substance or to any of the excipients

Ages: 21 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To assess the tolerability of quinagolide 200 μg/day in a dose-titration regimen in oocyte donors undergoing controlled ovarian hyperstimulation and at risk of developing OHSS | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad, Valencia, Spain